CLINICAL TRIAL: NCT05363904
Title: Environmental Impact and Immune Responses in Atopic Dermatitis Patients in Central Europe and Sub-Saharan Africa: A Prospective Study
Brief Title: Atopic Dermatitis: Sub-Saharan Africa vs. Central Europe
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Regional Dermatology Training Centre (RDTC), Moshi, Tanzania (Unknown); University Hospital Joseph Raseta Befelatanana in Antananarivo, Madagascar (Unknown)
Responsible Party: Principal Investigator, Marie-Charlotte Brüggen, Principal Investigator, University of Zurich
Other Study IDs: 2021-01869
Record Dates: First submitted 2022-03-04; First posted 2022-05-06 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples
  * Skin biopsies
  * Skin swabs
  * Nasal swabs
  * Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Atopic Dermatitis (Europe)
  Interventions: Other: Observation
- Healthy Controls (Europe)
  Interventions: Other: Observation
- Atopic Dermatitis (Tanzania)
  Interventions: Other: Observation
- Healthy Controls (Tanzania)
  Interventions: Other: Observation
- Atopic Dermatitis (Madagascar)
  Interventions: Other: Observation
- Healthy Controls (Madagascar)
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Questionnaires, Clinical Scores, Biomaterial Sampling

SUMMARY:
Many people are affected by atopic dermatitis (AD) worldwide. However, clinical studies on AD in Sub-Saharan Africa are rare and there is a lack of knowledge about possible differences in pathogenesis between European and African AD.

This study will collect clinical and laboratory data with the aim to compare clinical characteristics and immune responses in AD patients in Sub-Saharan Africa and Central Europe. Furthermore, relevant allergens as well as the nasal, skin and gut micro- and mycobiome will be investigated.

DETAILED DESCRIPTION:
Objectives of the project: Compare the following aspects in patients suffering from atopic dermatitis (AD) and healthy control (HC) participants in Central Europe (CE) vs. Sub-Saharan Africa (SsA):

* Clinical characteristics, life quality, treatments, and family history
* Immune mapping and barrier characterization of lesional and non-lesional skin
* Exploration of the serological and cutaneous immune signatures
* Investigation of the skin, nasal and gut microbiome (including bacteria and fungi)
* Comparison of the sensitization patterns and putting it into clinical context (food questionnaire, anamnesis about allergic symptoms, analysis of IgE and IgG levels)

ELIGIBILITY:
Inclusion Criteria:

AD patients:

* Age: ≥18 years
* Written informed consent given after information about the research project
* Suffering from active atopic dermatitis
* No active skin disease other than atopic dermatitis
* No known active inflammatory disease other than atopic dermatitis/atopic diseases

HC participants:

* Age: ≥18 years
* Written informed consent given after information about the research project
* No active skin disease
* No known atopic disease (atopic dermatitis, asthma, allergy, allergic rhinoconjuncitivitis)
* No known active inflammatory disease

Exclusion Criteria:

* Known or suspected systemic immunosuppression because of disease
* Systemic immunomodulatory/-suppressive treatment

  * Glucocorticoids or immunosuppressants (last 4 weeks) or
  * JAK inhibitors (last week) or
  * Omalizumab (last 4 weeks) or
  * Other biologicals e.g. dupilumab (last 2 months)
* Clinical signs of active bacterial, fungal or viral infection
* Systemic antibiotic, antimycotic or antiviral treatment 4 weeks prior to start
* Phototherapy 4 weeks prior to start
* Active neoplasia
* Undergoing surgery in the last 2 months
* Infarction (e.g. stroke), embolism, or thrombosis in the last 2 months
* Inability to follow the study procedures e.g. due to language problems, dementia etc. of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with active atopic dermatitis and healthy control participants
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Total and specific IgE and IgG levels | Day 0
  Will be put into clinical context with a questionnaire about food intake and allergic symptoms
Questionnaire about food intake | Day 0
  Information about how often the participants are consuming certain foods
Questionnaire about the presence of allergic symptoms | Day 0
  Information about symptoms upon allergen exposure
Description of clinical appearance of AD on black vs. white skin | Day 0
  Appearance, severity and distribution of the skin lesions
Stigmata of atopic constitution | Day 0
  The presence of atopic stigmata will be clinically assessed by study doctors by using a structured form
Skin microbiome (microbial colonization of the skin) | Day 0
  * Skin swabs will be taken at the following localizations: Antecubital crease, glabella, vertex, dorsal neck and lesional skin site
  * Analysis by isolation and sequencing of the microbial DNA
Change of the skin microbiome components over time | Day 0 and day 28
  * Skin swabs will be taken at the following localizations: Antecubital crease, glabella, vertex, dorsal neck and lesional skin site
  * Analysis by isolation and sequencing of the microbial DNA
Nasal microbiome (microbial colonization of the nasal vestibule) | Day 0
  * A nasal swab will be taken upon day 0
  * It will be used to grow cultures and analyse the microbial DNA
Gut microbiome (microbial colonization of the gut) | Day 0
  Analysis by isolation and sequencing of the microbial DNA
Cutaneous immune response | Day 0
  * Skin biopsies are optional and will be taken from lesional and non-lesional skin
  * They will be analyzed by imaging mass cytometry and spatial gene expression analysis
Systemic immune response | Day 0
  Olink multiplex proteomics analyses and characterization of PBMCs will be performed
Change of molecular and cellular mediators of the systemic immune response over time | Day 0 and day 28
  Olink multiplex proteomics analyses and characterization of PBMCs will be performed
Barrier dysfunction of the skin (Imaging Mass Cytometry) | Day 0
  Skin biopsies are optional and will be taken from lesional and non-lesional skin
Barrier dysfunction of the skin (Spatial gene expression analysis) | Day 0
  Skin biopsies are optional and will be taken from lesional and non-lesional skin
Family history of atopic diseases | Day 0
  - Assessment of whether parents, siblings or other family members suffer from atopic diseases
Questionnaire about current treatments | Day 0
  Participants will be asked about their intake of medication and their use of topical treatments
Life Quality measured by Dermatology Life Quality Index (DLQI) | Day 0
  * Min. 0, max. 30 points
  * Higher scores indicate a lower quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Charlotte Brüggen, Prof., Principal Investigator — University of Zurich; Daudi Mavura, Prof., Principal Investigator — RDTC Moshi; John Masenga, Prof., Principal Investigator — RDTC Moshi; Fandresena Sendrasoa, Dr., Principal Investigator — University Hospital Joseph Raseta Befelatanana
Locations (3):
- University Hospital Joseph Raseta Befelatanana, Antananarivo, Madagascar
- University Hospital Zurich, Zurich, Switzerland
- Regional Dermatology Training Centre (RDTC), Moshi, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fehr D, Lang C, Masenga J, Mavura D, Schmid-Grendelmeier P, Bruggen MC. Atopic dermatitis: The importance of future research in Africa. Allergy. 2023 Jan;78(1):327-328. doi: 10.1111/all.15422. Epub 2022 Dec 5. No abstract available. PMID 36468335
- See also: Flyer (University Hospital Zurich) — https://www.usz.ch/studie/neurodermitis-neurodermitis-in-europa-und-subsahara-afrika/